CLINICAL TRIAL: NCT00530361
Title: A Double-Blind, Randomized, Placebo-Controlled Study of Nesiritide Administered After Induction of Anesthesia in Heart Failure Patients With Renal Insufficiency Undergoing Coronary Artery Bypass Graft Surgery Requiring Cardiopulmonary Bypass (NAPA-CS)
Brief Title: An Efficacy and Safety Study for Nesiritide in Heart Failure Patients With Reduced Kidney Function Undergoing Coronary Artery Bypass Graft Surgery Requiring Cardiopulmonary Bypass (CPB Pump or Heart Lung Machine)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was withdrawn prior to patient dosing based on a business decision.
Sponsor: Scios, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR014266
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2011-07

CONDITIONS: Coronary Artery Bypass Surgery; Coronary Heart Disease; Coronary Artery Bypass Grafting; Cardiopulmonary Bypass; Ischemic Heart Disease; Heart Failure, Congestive
Keywords: Myocardial Ischemia; Kidney failure; CABG; Cardiopulmonary bypass (CPB) pump; Coronary Artery Bypass Surgery; Heart surgery; Nesiritide; Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease; Myocardial Ischemia; Heart Failure; Renal Insufficiency | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nesiritide

SUMMARY:
The purpose of this study is to assess whether nesiritide compared to placebo when given with standard of care therapies, helps preserve kidney function in heart failure (HF) patients undergoing heart bypass graft surgery that requires the use of a cardiopulmonary bypass machine (CPB pump or heart-lung machine).

DETAILED DESCRIPTION:
In coronary heart disease (CHD), the coronary arteries become clogged with calcium and fatty deposits. The deposits, called plaques, narrow the arteries that carry blood to the heart muscle and could cause ischemic heart disease (too little blood and oxygen reaching the heart muscle). Coronary Artery Bypass Graft (CABG) surgery is a treatment option for ischemic heart disease. CABG surgery is surgery to create new routes for blood to flow around narrowed and blocked arteries so that the heart muscle will receive needed oxygen and nutrients. Acute kidney injury is a serious risk of CABG surgery while on CPB pump (heart-lung machine), which could result from ischemia during and following surgery. This study is a double-blind (neither the patient or the doctor knows whether the patient is assigned to receive study drug or placebo), randomized (assigned to treatment by chance), placebo-controlled (study drug results compared to placebo results) study to determine the effectiveness of nesiritide compared to placebo when given to HF patients undergoing CABG surgery requiring the use of a CPB pump . The study drug (nesiritide) or placebo dose being studied is 0.010 mcg/kg/min via continuous IV infusion. The study hypothesis is that compared to placebo, nesiritide will reduce kidney ischemia, preserve glomerular filtration rate (GFR),which measures the rate at which the kidneys filter blood, and the need for dialysis or occurrence of death in HF patients who have undergone heart bypass surgery requiring the use of a cardiopulmonary bypass machine. Safety will be assessed through the collection of adverse events, clinical laboratory tests, vital signs, physical examinations and electrocardiograms at various time points throughout the study. The patients assigned to the nesiritide group will receive a continuous I.V. infusion at 0.010 mcg/kg/min of nesiritide for at least 48 hours and could be extended to up to 96 hours. The patients assigned to the placebo group will receive matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of congestive heart failure
* Documentation of left ventricular ejection fraction (LVEF)<= 40% within 90 days before surgery
* Pre-existing renal insufficiency with a glomerular filtration rate of <= 60 mL/min/1.73 m2 measured within 24 hours before surgery
* Scheduled to undergo coronary artery bypass graft (CABG) surgery with or without mitral valve replacement or repair on Cardiopulmonary Bypass machine.

Exclusion Criteria:

* History of cardiac disease or conditions in which cardiac output is dependent on venous return or Pulmonary disease (COPD), asthma, or other conditions that have required inpatient medical or surgical treatment within 60 days before surgery
* Documented systemic bacterial/fungal/viral infection within 72 hours before surgery
* Known acute renal failure or ongoing chronic dialysis at baseline
* Any of the following: mean pulmonary artery pressure <= 15 mmHg, central venous pressure < 6 mmHg, or systolic blood pressure < 90 mmHg before surgery
* Planned aortic valve repair or replacement
* Pregnant, suspected to be pregnant, or breast feeding
* Received an experimental drug or used an experimental medical device within 30 days before the planned start of study drug
* Known allergic reaction or sensitively to nesiritide or excipients
* Received commercial nesiritide within 48 hours before the planned start of study drug or was previously randomized in the NAPA-CS study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
The composite of a 25% decrease in postoperative glomerular filtration rate, occurrence of postoperative dialysis, and all-cause mortality through Day 30; The composite of occurrence of postoperative dialysis and all-cause mortality through Day 90.

SECONDARY OUTCOMES:
The occurrence of new-onset postoperative atrial fibrillation through 96 hours after randomization. The composite of re-intubation for respiratory failure and all-cause mortality through 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.